CLINICAL TRIAL: NCT04189289
Title: Comparison of the Efficacy of Ultrasound-guided Erector Spinae Plane Block for Postoperative Analgesia in Patients Undergoing Laparoscopic Bariatric Surgery
Brief Title: Laparoscopic Bariatric Surgery and Erector Spinae Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21/16
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2019-12

CONDITIONS: Obesity; Postoperative Pain; Bariatric Surgery
Keywords: Erector spinae plane (ESP) block; Laparoscopic bariatric surgery; Obesity; Postoperative pain
MeSH Terms: conditions — Obesity; Pain, Postoperative; Bites and Stings | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomised controlled
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP block group (Active Comparator): Before anaesthesia induction; bilateral ESP block will be performed under the guidance of USG. Patients will be administered paracetamol 1 gr IV every 8 hours in the postoperative period. Standardized postoperative tramadol i.v. patient controlled analgesia (PCA) protocol will be performed (3 mg/ml, total volume 100 ml, 10 mg bolus dose, 20 min locked period, without continuous delivery, no basal infusion).
  Interventions: Procedure: ESP block group
- Control group (Sham Comparator): Patients will be administered paracetamol 1 gr IV every 8 hours in the postoperative period. Standardized postoperative tramadol i.v. PCA analgesia protocol will be performed (3 mg/ml, total volume 100 ml, 10 mg bolus dose, 20 min locked period, without continuous delivery, no basal infusion).
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: ESP block group — USG probe will be placed in a longitudinal parasagittal orientation 3 cm lateral to T7 spinous process. The erector spinae muscles will be identified hyperechoic transverse process. The patient's skin will be anesthetized with 2% lidocaine. A 21-gauge 10-cm needle was inserted using an in-plane superior-to-inferior approach or an out-plane approach. Following confirmation of the correct position of the needle with 5 ml normal saline, a dose of 20 ml %0.25 bupivacaine will be administered. The same procedure will be performed at the other site (totally 40 ml %0.25 bupivacaine). Standard pain follow up and monitorization will be performed.
  Arms: ESP block group
Procedure: Control group — The patients in this group will be performed no block. Standard pain follow up and monitorization will be performed.
  Arms: Control group

SUMMARY:
The aim of the study is to evaluate the effect of erector spinae plane (ESP) block on postoperative analgesic consumption in patients undergoing laparoscopic bariatric surgery

DETAILED DESCRIPTION:
Laparoscopic sleeve gastrectomy is one of the most common surgical procedure that is chosen for bariatric surgery. Postoperative pain after bariatric surgery can de significant. Narcotic analgesics are often used to manage the postoperative pain in patients undergoing bariatric surgery. However, these drugs causes many undesirable adverse effects such as nausea, constipation, and respiratory depression.

The ultrasound (USG) guided ESP block was first defined in 2016. With the administration of local anesthesia between the transverse process of the vertebra and the erector spinae muscle, it is stated that the effect mechanism of ESP is that spread blocks the ventral and dorsal rami to the paravertebral area. In the literature, it has been shown that bilateral USG guided ESP block provides effective analgesia after bariatric surgery.

The aim of the study is to evaluate the effect of ESP block on postoperative analgesic consumption in patients undergoing laparoscopic bariatric surgery

ELIGIBILITY:
Inclusion Criteria:

* elective bariatric surgery
* American Society of Anesthesiology (ASA) II-III
* 18 - 65 years
* body mass index (BMI) 40-60 kg/m2

Exclusion Criteria:

* ASA ≥4
* under 18 years of age or over 65 years of age
* declining to give written informed consent
* have neurological and/or psychiatric disorders
* cooperation cannot be established
* accompanying laparoscopic cholecystectomy or paraumbilical hernia repair
* history of bariatric surgery
* the block cannot be applied due to bleeding disorders or localized skin infection at the injection site
* with hepatic, neuromuscular, cardiac and/or renal failure
* history of allergy to the local anesthetics
* patients undergoing open surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-06 (Actual)

PRIMARY OUTCOMES:
analgesia consumption | 24 hours
  postoperative 24 hours

SECONDARY OUTCOMES:
Postoperative Numeric Rating Scale (NRS) score | postoperative 0, 1, 3, 6, 12, 24 hours
  postoperative pain assessment will be performed using NRS score (NRS 0=no pain, NRS 10= most severe possible).

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Karaveli, Principal Investigator — Antalya TRH
Locations (1):
- Antalya Training and Research Hospital, Department of Anesthesiology and Reanimation, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chin KJ, Malhas L, Perlas A. The Erector Spinae Plane Block Provides Visceral Abdominal Analgesia in Bariatric Surgery: A Report of 3 Cases. Reg Anesth Pain Med. 2017 May/Jun;42(3):372-376. doi: 10.1097/AAP.0000000000000581. PMID 28272292
- [Background] Tulgar S, Kapakli MS, Senturk O, Selvi O, Serifsoy TE, Ozer Z. Evaluation of ultrasound-guided erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy: A prospective, randomized, controlled clinical trial. J Clin Anesth. 2018 Sep;49:101-106. doi: 10.1016/j.jclinane.2018.06.019. Epub 2018 Jun 15. PMID 29913392